CLINICAL TRIAL: NCT06730646
Title: Testing Different Anti-smoking Messages Among Chinese Young Adult Smokers and Nonsmokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Di Pei, Postdoctoral Research Associate, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H24245
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Smoking Prevention
Keywords: anti-smoking; health communication; smoking behavior
MeSH Terms: conditions — Smoking | interventions — Tobacco Smoke Pollution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Health effects (Experimental): Participants will receive messages with information about smoking-related diseases.
  Interventions: Behavioral: Health effects
- Tobacco industry manipulation (Experimental): Participants will receive messages with information about how the tobacco industry uses targeted marketing and manipulative tactics aimed at youth and young adults.
  Interventions: Behavioral: Tobacco industry manipulation
- Secondhand smoke (Experimental): Participants will receive messages with information about secondhand smoke exposure.
  Interventions: Behavioral: Secondhand smoke
- Mental Health (Experimental): Participants will receive messages with information about the effects of smoking on mental health.
  Interventions: Behavioral: Mentral health
- Social acceptability (Experimental): Participants will receive messages that portray smoking as socially unacceptable in China.
  Interventions: Behavioral: Social acceptability
- Control (Other): Participants will receive messages about bottled water which should have no impact on the outcomes of interest.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Health effects — Participants in this arm will watch 3 short videos about the smoking-related diseases during the survey data collection.
  Arms: Health effects
Behavioral: Tobacco industry manipulation — Participants in this arm will watch 3 short videos about how the tobacco industry uses targeted marketing and manipulative tactics aimed at youth and young adults during the survey data collection.
  Arms: Tobacco industry manipulation
Behavioral: Secondhand smoke — Participants in this arm will watch 3 short videos about the risks of secondhand smoke exposure during the survey data collection.
  Arms: Secondhand smoke
Behavioral: Mentral health — Participants in this arm will watch 3 short videos about the effects of smoking on mental health during the survey data collection.
  Arms: Mental Health
Behavioral: Social acceptability — Participants in this arm will watch 3 short videos about how smoking is socially unacceptable in China during the survey data collection.
  Arms: Social acceptability
Behavioral: Control — Participants in this arm will watch 3 short videos about drinking bottled water during the survey data collection. These messages display specific water products and describe hydration as a healthy activity.
  Arms: Control

SUMMARY:
Young adults are particularly vulnerable to psychological distress during the transition from adolescence to adulthood, making them more susceptible to developing persistent substance use. The tobacco industry capitalizes on this vulnerability by using marketing tactics to promote tobacco initiation and facilitate the progression from experimental tobacco use to long-term use. In China, where the average age of starting daily smoking is 21.1 years old, the number of current young adult smokers exceeds 29 million. It is crucial to develop effective communication messages to counter the tobacco industry's marketing strategies and protect the health of young adults in China. This project aims to test the effects of different anti-smoking message themes among Chinese young adults. In this online randomized clinical trial, participants will be randomly assigned to one of five antismoking message conditions. The investigators will compare the effects of these themes with each other and with the control condition.

DETAILED DESCRIPTION:
In this study, the investigators will examine the effectiveness of different anti-smoking themes in reducing intention to smoke among Chines young adults. The study will recruit 1500 adults aged 18-25 years old, including 750 current smokers and 750 non-smokers, evenly split between male and female.

The study will be conducted through a self-administered, web-assisted online survey software. Participants will be asked to consent to participate in this study via a consent form presented at the beginning of the survey. Consented participants will be randomized to one of six conditions (each represents a level of the independent variable: anti-smoking message theme): 1) Health effects 2) Tobacco industry manipulation 3) Mental health 4) Secondhand smoke 5) Social acceptability 6) Control messages with no cigarette-related content.

The study has two sessions. In session 1, participants will complete a 20-minute survey. The survey will begin with questions assessing demographic characteristics. Then participants will be shown intervention or control messages (watch three 30-second video in each condition), and beliefs and future intention to smoke cigarettes will be assessed.

Two weeks after session 1, participants will be asked to complete a 5-minute survey in session 2 of the study. The survey will measure participants' recall of the messages and smoking behaviors in the past two weeks after message exposure.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 18-25 years old

  * Current residency in China
  * Current smokers - having smoked at least 100 cigarettes in a lifetime and currently smoking every day or some days
  * Nonsmokers - having not smoked 100 cigarettes in a lifetime and do not currently smoke cigarettes
  * Can to read, speak, and understand Mandarin Chinese

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1541 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Intention to use tobacco | Immediately after message exposure
  A five-item scale measuring future intentions to smoke cigarettes and other forms of tobacco over the next year.
  Response options: from 1 (very unlikely) to 5 (very likely).
  Higher scores represent stronger intention to use tobacco.

SECONDARY OUTCOMES:
Perceived harm of smoking | Immediately after message exposure
  Measured with a single item, assesses participant's perception of own risk of overall harm to health under conditions of smoking every day. Response options range from 1 (Not at all likely) to 5 (Extremely likely), with higher scores representing a better outcome.
Perceived Message Effectiveness | Immediately after message exposure
  A three-item scale measuring to what extent participants think the messages they saw discourage them from wanting to smoke, make smoking seem unpleasant, and make them concerned about health risks of smoking.
  Response options: from 1 (Disagree) to 4 (Neither Disagree nor Agree) to 7 (Strongly Agree).
  Higher scores represent a better outcome. The final perceived message effectiveness score is the mean of the response to the three items.
Quit intention | Immediately after message exposure
  Only measured among smokers. A two-item scale measuring to what extent participants are interested in quitting in the next 6 month. Response options are from 1 (Not at all likely) to 5 (Extremely likely), with higher scores representing a better outcome. The final quit intention score is the mean of the response to the two items.
Smoking behavior | Two weeks after message exposure
  Single item measuring the average number of cigarettes smoked per day in the past two weeks.
Intention to use tobacco in follow-up test | Two weeks after message exposure
  A five-item scale measuring future intentions to smoke cigarettes and other forms of tobacco over the next year. Response options: from 1 (very unlikely) to 5 (very likely). Higher scores represent stronger intention to use tobacco.

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia State university, Atlanta, Georgia, United States
- Online, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No